CLINICAL TRIAL: NCT07086157
Title: Effects of Low-FODMAP Diet and Probiotics on Gastrointestinal Symptoms, Behavior Problems, and Microbiota in Children With Autism Spectrum Disorder and Gastrointestinal Symptoms
Brief Title: Low-FODMAP Diet and Probiotics: Effects on Gut, Behavior, and Microbiota in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Collaborators: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Pınar Polat, Doctor Dietitian, Marmara University Pendik Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2023.1132
Record Dates: First submitted 2025-07-05; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder; Functional Gastrointestinal Disorders
Keywords: autism spectrum disorder; probiotics; gut microbiota; low FODMAP diet; gastrointestinal symptoms
MeSH Terms: conditions — Autism Spectrum Disorder; Gastrointestinal Diseases | interventions — Probiotics; FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-FODMAP Diet + Probiotic Supplement (Experimental): Participants in this arm received the same probiotic supplement as the other group once daily for 4 weeks, in combination with a personalized low-FODMAP diet. The diet was planned and monitored by a registered dietitian to ensure compliance and nutritional adequacy.
  Interventions: Dietary Supplement: Probiotic; Other: Low-FODMAP Diet
- Probiotic Supplement Only (Experimental): Participants in this arm received a multi-strain probiotic supplement containing four bacterial strains (Lactobacillus acidophilus L1, Bifidobacterium longum LBL-01, Lactobacillus rhamnosus, and Saccharomyces boulardii) once daily for 4 weeks. No dietary restrictions or modifications were applied in this group.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — A probiotic supplement in capsule form containing 4 strains of microorganisms, with a total of 10 × 10⁹ CFU (colony-forming units) per capsule. The strain composition per capsule was:
  Lactobacillus acidophilus L1 - 2.9 × 10⁹ CFU, Bifidobacterium longum LBL-01 - 2.9 × 10⁹ CFU, Lactobacillus rhamnosus - 2.9 × 10⁹ CFU, Saccharomyces boulardii - 1.3 × 10⁹ CFU. Each participant in this arm took one capsule per day in the morning on a full stomach, for a duration of 4 weeks. No other dietary interventions were applied to this group. This probiotic supplement was chosen because the strains in its content are among the most frequently researched and known strains in terms of intestinal health. Additionally, it does not contain FOS or inulin due to FODMAP restriction.
  .
Other: Low-FODMAP Diet — A structured low-FODMAP diet intervention designed to restrict intake of fermentable oligosaccharides, disaccharides, monosaccharides, and polyols. The diet was individualized and monitored by a registered dietitian over a 4-week period to ensure adherence and nutritional adequacy.
  Arms: Low-FODMAP Diet + Probiotic Supplement

SUMMARY:
The goal of this clinical trial was to evaluate whether a low-FODMAP diet and probiotic supplements could reduce gastrointestinal (GI) symptoms and behavior problems in children with autism spectrum disorder (ASD) who also experienced GI issues. The main questions it aimed to answer were:

Did a low-FODMAP diet and/or probiotics improve GI symptoms such as constipation, diarrhea, and abdominal pain?

Did these interventions help reduce behavior problems such as irritability, lethargy, stereotypy, hyperactivity, and speech disorder ?

Researchers compared two groups:

1. Children who received a daily probiotic supplement containing 4 strains for 4 weeks
2. Children who received both the probiotic supplement and followed a low-FODMAP diet

This comparison aimed to determine whether the combination of diet and probiotics had greater benefits than probiotics alone.

Participants:

Took the assigned intervention(s) for 4 weeks

Provided stool samples for gut microbiota analysis

Completed assessments of GI symptoms and behavior using validated questionnaires

DETAILED DESCRIPTION:
This randomized, controlled, parallel-group clinical trial aimed to investigate the effects of a low-FODMAP diet and multi-strain probiotic supplementation on gastrointestinal (GI) symptoms, behavioral problems, and gut microbiota composition in children with Autism Spectrum Disorder (ASD) who presented with concurrent GI complaints.

Children aged 6 to 12 years with clinically diagnosed ASD and GI symptoms were recruited. A total of 16 participants were randomly assigned into two equal groups (n=8 per group). One group received a probiotic supplement containing four bacterial strains daily for 4 weeks, while the second group received the same probiotic supplement in combination with a low-FODMAP diet over the same period. The randomization was stratified and allocation was blinded to the data analysts.

Interventions Probiotic group: A commercially available probiotic blend (containing Lactobacillus acidophilus, Bifidobacterium longum, Lactobacillus rhamnosus, and Saccharomyces boulardii) was administered once daily for 4 weeks.

Low-FODMAP + Probiotic group: In addition to the probiotic supplement, participants received individualized nutrition counseling and followed a standardized low-FODMAP diet protocol under dietitian supervision for 4 weeks.

Data Collection and Measures GI symptoms were assessed using the Pediatric Gastrointestinal Symptoms Questionnaire - Rome III Version (QPGS-RIII) and the Bristol Stool Scale (BSS).

Behavioral outcomes were evaluated using the Aberrant Behavior Checklist (ABC), focusing on subscales including irritability, lethargy-social withdrawal, stereotypy, hyperactivity, and inappropriate speech.

Dietary intake was recorded using 3-day food diaries to determine intake of daily FODMAP amount.

Microbiota composition was analyzed from fecal samples using 16S rRNA gene sequencing and LEfSe (Linear Discriminant Analysis Effect Size) for taxonomic biomarker discovery.

Quality Control and Data Validation All participants were monitored weekly to ensure adherence to interventions and assess adverse effects.

Dietary intake data were validated against food portion models and caregiver interviews.

Stool sample processing followed standardized protocols: DNA was extracted, amplified, and sequenced using Illumina platforms.

A pre-defined bioinformatics pipeline was used for quality filtering, taxonomic assignment, and alpha/beta diversity analysis.

Internal consistency checks and double data entry validation were applied to all behavioral and symptom questionnaires.

Statistical Analysis Statistical analysis was performed using SPSS v25 and R. Paired and independent-sample t-tests or Wilcoxon signed-rank tests were applied based on distribution normality. Microbiota diversity indices (Shannon, Simpson, Chao1) and taxonomic differences were compared across groups and time points. Spearman correlation analyses were used to explore associations between microbiota shifts and clinical parameters. A p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Autism Spectrum Disorder by a specialist at Marmara University Pendik Training and Research Hospital Child and Adolescent Psychiatry Clinic
* Aged between 6 and 12 years
* Diagnosed with functional gastrointestinal symptoms according to Rome IV criteria
* Willing to participate by signing informed consent and assent forms (by both child and parent)

Exclusion Criteria:

* Following any other dietary intervention at the time of study initiation
* Routine use of prebiotics or probiotics
* Use of antibiotics within the 4 weeks prior to the study
* Presence of active diarrhea due to intestinal infection or similar condition
* Diagnosis of other gastrointestinal diseases besides functional GI symptoms

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Aberrant Behavior Checklist (ABC) Irritability Subscale Score | Baseline and after 4 weeks of intervention
  Change in caregiver-reported irritability scores as measured by the Aberrant Behavior Checklist Irritability Subscale, a standardized behavioral rating scale.
Change in Aberrant Behavior Checklist (ABC) Hyperactivity Subscale Score | Baseline and after 4 weeks of intervention
  Change in hyperactivity scores, as assessed by the caregiver-completed Hyperactivity Subscale of the Aberrant Behavior Checklist (ABC), a standardized behavioral rating scale.
Change in Aberrant Behavior Checklist (ABC) Lethargy-Social Withdrawal Subscale Score | Baseline and after 4 weeks of intervention
  Change in lethargy-social withdrawal scores, as assessed by the caregiver-completed Lethargy-Social Withdrawal Subscale of the Aberrant Behavior Checklist (ABC), a standardized behavioral rating scale.
Change in Aberrant Behavior Checklist (ABC) Stereotypy Subscale Score | Baseline and after 4 weeks of intervention
  Change in stereotypy scores, as assessed by the caregiver-completed Stereotypy Subscale of the Aberrant Behavior Checklist (ABC), a standardized behavioral rating scale.
Change in Aberrant Behavior Checklist (ABC) Inappropriate Speech Subscale Score | Baseline and after 4 weeks of intervention
  Change in inappropriate speech scores, as assessed by the caregiver-completed Inappropriate Speech Subscale of the Aberrant Behavior Checklist (ABC), a standardized behavioral rating scale.
Change in Presence of Functional Gastrointestinal Symptoms as Measured by the QPGS-RIII | Baseline and after 4 weeks of intervention
  Change in the presence of any functional gastrointestinal symptoms as determined by caregiver responses to the Pediatric Gastrointestinal Symptoms Questionnaire - Rome III (QPGS-RIII), a validated diagnostic tool for functional gastrointestinal disorders in children.

SECONDARY OUTCOMES:
Change in Gut Microbiota Alpha Diversity (Shannon Index) | Baseline and after 4 weeks of intervention
  Change in microbial alpha diversity of stool samples, assessed using 16S rRNA gene sequencing and expressed as the Shannon diversity index.
Change in Gut Microbiota Beta Diversity (UniFrac Analysis) | Baseline and after 4 weeks of intervention
  Change in microbial beta diversity of stool samples, assessed using 16S rRNA gene sequencing and analyzed with UniFrac distance metrics to evaluate differences in microbial community composition between samples.
Change in Relative Abundance of Specific Bacterial Genera | Baseline and after 4 weeks of intervention
  Change in the relative abundance (%) of key bacterial genera identified through 16S rRNA sequencing and LEfSe analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Polat, PhD, Principal Investigator — Marmara University Pendik Training and Research Hospital; Neşe Perdahlı Fiş, Prof Dr, Study Chair — Marmara University Pendik Training and Research Hospital; Özlem Aytekin, AProf Dr, Study Director — Saglik Bilimleri Universitesi; Fatih Özbey, Prof Dr, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Marmara Univesity Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 2 years after the publication of results.
Access Criteria: Individual participant data (IPD), including raw sequence data, will be shared with qualified researchers upon reasonable request. Raw 16S rRNA sequencing data are publicly available through the National Library of Medicine's Sequence Read Archive (SRA) under accession number [PRJNA1112427]. Other IPD can be requested for methodologically sound research purposes by submitting a proposal to the principal investigator. Requests will be reviewed for scientific validity and ethical compliance. Data will be shared via secure transfer after approval and signing a data use agreement.
URL: https://www.ncbi.nlm.nih.gov/sra

REFERENCES:
- [Background] Lee JC, Chen CM, Sun CK, Tsai IT, Cheng YS, Chiu HJ, Wang MY, Tang YH, Hung KC. The therapeutic effects of probiotics on core and associated behavioral symptoms of autism spectrum disorders: a systematic review and meta-analysis. Child Adolesc Psychiatry Ment Health. 2024 Dec 19;18(1):161. doi: 10.1186/s13034-024-00848-3. PMID 39702309
- [Background] Iglesias-Vazquez L, Van Ginkel Riba G, Arija V, Canals J. Composition of Gut Microbiota in Children with Autism Spectrum Disorder: A Systematic Review and Meta-Analysis. Nutrients. 2020 Mar 17;12(3):792. doi: 10.3390/nu12030792. PMID 32192218
- [Background] Srikantha P, Mohajeri MH. The Possible Role of the Microbiota-Gut-Brain-Axis in Autism Spectrum Disorder. Int J Mol Sci. 2019 Apr 29;20(9):2115. doi: 10.3390/ijms20092115. PMID 31035684
- [Background] Settanni CR, Bibbo S, Ianiro G, Rinninella E, Cintoni M, Mele MC, Cammarota G, Gasbarrini A. Gastrointestinal involvement of autism spectrum disorder: focus on gut microbiota. Expert Rev Gastroenterol Hepatol. 2021 Jun;15(6):599-622. doi: 10.1080/17474124.2021.1869938. Epub 2021 Jan 5. PMID 33356668
- [Background] Socala K, Doboszewska U, Szopa A, Serefko A, Wlodarczyk M, Zielinska A, Poleszak E, Fichna J, Wlaz P. The role of microbiota-gut-brain axis in neuropsychiatric and neurological disorders. Pharmacol Res. 2021 Oct;172:105840. doi: 10.1016/j.phrs.2021.105840. Epub 2021 Aug 24. PMID 34450312
- [Background] Martinez-Gonzalez AE, Andreo-Martinez P. The Role of Gut Microbiota in Gastrointestinal Symptoms of Children with ASD. Medicina (Kaunas). 2019 Jul 26;55(8):408. doi: 10.3390/medicina55080408. PMID 31357482
- [Background] Leader G, Abberton C, Cunningham S, Gilmartin K, Grudzien M, Higgins E, Joshi L, Whelan S, Mannion A. Gastrointestinal Symptoms in Autism Spectrum Disorder: A Systematic Review. Nutrients. 2022 Apr 1;14(7):1471. doi: 10.3390/nu14071471. PMID 35406084
- See also: Full-text thesis record in the Turkish National Thesis Center. The thesis no is 888255. — https://tez.yok.gov.tr/UlusalTezMerkezi/
- Available data/document: Individual Participant Data Set: PRJNA1112427 — https://www.ncbi.nlm.nih.gov/sra — Raw 16S rRNA sequencing data are publicly available through the National Library of Medicine's Sequence Read Archive (SRA) under accession number PRJNA1112427.